CLINICAL TRIAL: NCT00173758
Title: The Expression of IL-15 and Its Receptor in Uterine NK Cells and Clinical Applications
Brief Title: The Expression of IL-15 and Its Receptor in Decidua
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9361701276
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-12-21 (Estimated); Status verified 2005-06

CONDITIONS: Pregnancy; Infertility
Keywords: IL-15; IL-15 receptor; decidual natural killer cells; endometrium
MeSH Terms: conditions — Infertility

INTERVENTIONS:
Procedure: co-culture of embryos and endometrial cells

SUMMARY:
Human decidual tissue appears to play an important role not only in nurturing the implanted embryos, but also in preventing its rejection by the maternal immune system. Insight into the maternal immunologic modulations during implantation is our main research interests. Our previous studies have shown that most lymphocytes in deciduae are natural killer cells. However, their phenotype is CD16-CD56+CD3-, which is different from that of peripheral natural killer cells. More importantly their cytotoxic activity is decreased and they can't attack the cytotrophoblasts. All of these contributes to no rejection developing at the fetomaternal interface and are related to success of pregnancy.

In 1994, a new cytokine IL-15 was first discovered, which could act on the IL-15 and IL-2 receptors to stimulate the activation and propagation of the lymphocytes. Let us want to study the critical role of IL-15 in the endometrial lymphocytes. In this study, we try to analyze the distribution of IL-15 and its receptor in deciduae. We will clarify whether the IL-15 receptor exists on the decidual natural killer cells and it is regulated by sexual hormones or not and whether their cytotoxic activity will change after IL-15 action. Furthermore, we will demonstrated whether the IL-15 receptor exists on the embryo cells and IL-15 might improve the quality of the embryo. We also design a co-culture system of the embryo and autologous endometrial cells to improve the success rate of in vitro fertilization.

DETAILED DESCRIPTION:
The expression of IL-15 and IL-15Rα in the lymphocytes of peripheral blood and decidua during early pregnancy

1. Collection of specimens Collect the peripheral blood and decidual tissue from 20-30 pregnant women of 6-8 weeks gestational age during D&C procedure due to multiparity.
2. Immunohistochemical stain of decidual tissue The frozen section of decidual tissue was performed according to recommended procedures. First antibody, mouse anti-human IL-15 or IL-15Rα monoclonal antibody, second antibody, peroxidase-labeled goat anti-mouse polyclonal antibody, and color reagents were added sequentially. Finally the slides were counter-stained with hematoxylin.
3. Separation of mononuclear cells Decidual tissue and peripheral blood samples were taken from each pregnant woman at the time of abortion. In order to minimize contamination by blood, the decidual tissue was macroscopically separated from the chorionic villi, washed twice with Hank's balanced salt solution, cut into small pieces, washed twice again, and passed through a 1.9-mm mesh to remove the residual blood without enzymatic treatment. These samples were then filtered through a 45.7-μm stainless steel mesh to remove tissue debris. The filtered solution was layered over a Ficoll-Paque PLUS gradient and centrifuged for 45 minutes at 400g. An enriched cell suspension of mononuclear cells was collected at the interface and then washed twice with RPMI-1640 medium. Peripheral blood mononuclear cells were also isolated by Ficoll-Paque PLUS sedimentation.
4. Cytometric analyses The expression of intracellular IL-15 and surface IL-15Rα in mononuclear cells were analyzed with flow cytometry. The antibody combinations included: FITC/PE/PerCP- CD4/IL-15/CD3, CD8/IL-15/CD3, CD56/IL-15/CD3, CD4/IL-15Rα/CD3, CD8/IL-15Rα/CD3, CD56/IL-15Rα/CD3.
5. Separation of CD4+ cells, CD8+ cells and NK cells The CD4+ cells, CD8+ cells and NK cells in peripheral blood and deciduae were separated respectively with magnetic activated cell sorter (MACS).
6. Real-time PCR of IL-15 and IL-15Rα mRNA The total RNA in CD4+ cells, CD8+ cells and NK cells was extracted with Trizol, and was transformed to cDNA with reverse transcription. Real-time PCR was performed using different probes for ß-actin, IL-15 and IL-15Rα with ABI PRISM 7700 Sequence Detector System. The primer sequences were: ß-actin, 5' GTG GGG CGC CCC AGG CAC CA; 5' CTC CTT AAT GTC ACG CAC GAT TTC; IL-15, 5' GGC TTT GAG TAA TGA GAA TTT CGA; 5' ATC AAT TGC AAT CAA GAA GTG TTG; IL-15Rα, 5' GGC GAC GCG GGG CAT CAC; 5' TCG CTG TGG CCC TGT GGA TA.
7. Functional tests of CD4+ cells, CD8+ cells and NK cells

   1. Proliferative assay Using incorporation of BrdU during cellular proliferation, the proliferative ability of CD4+ cells, CD8+ cells and NK cells was assessed when different concentrations of IL-15 and IL-2 were added.
   2. Secretion assay The concentrations of IFN-γ, IL-6 and IL-10 in the supernatant were detected using ELISA kits when different concentrations of IL-15 and IL-2 were added into the culture medium.
   3. Fluoresence-based cellular cytotoxicity- FCC assay NK- and CTL-mediated cytolysis of target cells constitutes a form of apoptosis, and is accompanied by many of the same events, including caspase activation. We incorporated the fluorogenic substrate for caspase 6 into the target cells (K562 cells and autologous cytotrophoblasts) and measured the caspase activation by detecting the fluorescence emitted from the cleaved substrate.

The expression of IL-15 and IL-15Rα in the human embryo before and after co-cultured with autologous endometrium

1. Immunocytochemical stain of human embryo Human embryos from IVF program were fixed on the adhesion slide with ice-cold Fixation Buffer. The phycoerythrin-conjugated anti-IL-15 monoclonal antibody or biotinylated anti-human IL-15Rα antibody and streptavidin- fluorescein isothiocyanate (SAv-FITC) Conjugate were added. The fluoroscope was used to detect the fluorescence emitted from the targets.
2. Single-cell PCR of IL-15 and IL-15Rα mRNA Using the principle of biotin/streptavidin "capture", the embryo mRNA was isolated with Micro RNA Isolation Kit, labeled with biotin-labeled oligo dT-probe and extracted with streptavidin-coated tubes. After transforming to cDNA, real-time PCR was performed using different probes for ß-actin, IL-15 and IL-15Rα with ABI PRISM 7700 Sequence Detector System, as described above.
3. Separation of autologous endometrial cells A luteal phase endometrial biopsy was performed in a cycle before the patient's IVF procedure with a Pipelle Endometrial Suction Curette. The tissue was digested with 0.2% collagenase type 2 and allowed to settle by differential sedimentation at unit gravity. The above steps were repeated four times and the supernatant was collected. After differential sedimentation at unit gravity, the supernatant, containing the stroma-enriched fraction, was transferred into tissue culture flasks for future use. The tissue pieces, which remained after the four digests, were resuspended in 10 mL HBSS. After approximately 30 seconds, the top 8 mL was allowed to settle at unit gravity. This sedimentation, containing glandular-enriched fraction, was resuspended in RPMI and plated into tissue culture flasks for future co-culture.
4. Autologous endometrial co-culture of human embryo Approximately an equal amount of the glandular and stromal cells were mixed on the estimated day before the administration of hCG during the patient's IVF cycle. About 3x10^5 cells were seeded into a four-well tissue culture plate and the zygotes were placed into the co-culture system or conventional medium (human tubal fluid plus 15% maternal serum). Cleavage rates and morphological appearance were assessed daily. The morphologically best embryos were transferred back to the patient 72 hours after retrieval irrespective of culture system. The implantation rate was defined as the number of intrauterine sacs with fetal cardiac activity per number of embryos transferred. Clinical pregnancies included only those pregnancies with a fetal heart beat documented on transvaginal ultrasound by day 49.
5. The cytokine distribution in co-culture medium The cytokines, including Th1 cytokines (IL-2 and IFN-γ), Th2 cytokines (IL-4, IL-6 and IL-10) and IL-15 were determined by ELISA technique in the co-culture medium before and after embryos plated.
6. Immunocytochemical stain of human endometrial glandular and stromal cells The purified endometrial glandular and stromal cells were washed twice with cold Wash Buffer to remove the cytokines adherent on the cells. These cells were then fixed on the adhesion slide with ice-cold Fixation Buffer. The phyco- erythrin-conjugated anti-IL-15 monoclonal antibody or biotinylated anti-human IL-15Rα antibody and streptavidin-fluorescein isothiocyanate (SAv-FITC) Conjugate were added. The fluoroscope was used to detect the fluorescence emitted from the targets.
7. Real-time PCR of IL-15 and IL-15Rα mRNA from human endometrial glandular and stromal cells The total RNA in endometrial glandular and stromal cells was extracted with Trizol, and transformed to cDNA with reverse transcription. Real-time PCR was performed using different probes for ß-actin, IL-15 and IL-15Rα with ABI PRISM 7700 Sequence Detector System, as described above.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 20 and 40 years
* Written informed consent
* Regular cycles, between 21 and 35 days, within the last 6 months before pregnancy
* Early pregnancy between 4 to 10 weeks of gestation

Exclusion Criteria:

* Abnormal vaginal bleeding
* Concomitant treatment with other drugs
* Autoimmune diseases
* Pelvic inflammation with last 3 months
* Having any associated malignancy
* Unable or unwilling to comply fully with the protocol

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2005-09

PRIMARY OUTCOMES:
Fertilization rate of oocytes
Implantation rate of embryos
Pregnancy rate

CONTACTS AND LOCATIONS:
Overall Officials: Kuang-Han Chao, M.D., Principal Investigator — Department of Obstetrics and Gynecology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan